CLINICAL TRIAL: NCT02206932
Title: An Open Label, Pilot Study to Investigate the Safety and Efficacy of 12 Weeks of Simeprevir and Sofosbuvir, for HIV-infected, HCV Genotype 1 Patients With Advanced Fibrosis
Brief Title: A Study of the Safety and Effectiveness of Simeprevir and Sofosbuvir for Patients With HIV and Hepatitis C
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: never opened
Sponsor: University of California, San Francisco (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC435HPC2008
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C, Chronic; HIV CDC Category A1
Keywords: Hepatitis C; HIV; Simeprevir; Sofosbuvir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sofosbuvir + Simeprevir (Other): Subjects will be enrolled and treated with simeprevir 150 mg and sofosbuvir 400 mg once daily for 12 weeks
  Interventions: Drug: Sofosbuvir + Simeprevir

INTERVENTIONS:
Drug: Sofosbuvir + Simeprevir
  Other Names: Sovaldi; Olysio; TMC435

SUMMARY:
This is a study of the safety and effectiveness of the hepatitis C medications sofosbuvir and simeprevir in patients who have both the HIV and hepatitis C (HCV) viruses.

DETAILED DESCRIPTION:
This is a research study of an investigational combination of two hepatitis C medications call sofosbuvir (SOF) and simeprevir (SMV). Both medications are approved by the U.S. Food and Drug Administration (FDA) for treatment of hepatitis C in combination with other medications. The combination sofosbuvir and simeprevir has not been approved by the FDA and is being tested as an investigational combination in research studies such as this. The purpose of this study is to see if SOF + SMV given for 12 weeks is safe and able to clear the Hepatitis C virus (HCV) from subjects who are co-infected with HIV-1 and who have scarring of the liver (fibrosis of 3 or 4 on a scale of 0-4, with 4 as the most scarring, also known as cirrhosis).

This study is an investigator-initiated clinical trial sponsored by University of California, San Francisco (UCSF), with support and the study drug simeprevir provided by Janssen Scientific Affairs, LLC.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or female, age ≥ 18 years
* Body mass index (BMI) ≥ 18 kg/m2
* HCV RNA ≥ 104 IU/mL at Screening
* HCV genotype 1 at screening or with prior documentation. Any non-definitive genotype results will exclude the subject from study participation
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
* Fibrosis determination: Fibrosis of Metavir F3/F4 may be established by one of the following:

  1. Liver biopsy at any point in time with Metavir score F3/F4, or equivalent on an alternative scale.
  2. Fibroscan ≥ 9.5 kPA
  3. FibroSURE: ≥ 0.58
* Liver imaging within 12 months prior to Baseline/Day 1 is required in subjects with known cirrhosis to exclude hepatocellular carcinoma (HCC). Acceptable liver imaging includes ultrasound, CT scan or MRI.
* HCV treatment status of one of the following:

  1. HCV Treatment-Naive: No prior exposure to any IFN, RBV, or other approved or experimental HCV-specific DAA agents
  2. HCV Treatment-Experienced: Virologic failure after treatment with PEG-IFN+RBVor standard IFN +RBV. Prior exposure to HCV polymerase or protease inhibitors is exclusionary. Prior treatment experienced patients will be categorized as one of the following:

  i. HCV Treatment-Intolerant: Subjects that discontinued HCV treatment due to development or significant worsening of a treatment related adverse event ii. Null responder: HCV RNA < 2 log10 decline during first 12 weeks of treatment iii. Partial responder: HCV RNA ≥ 2 log10 decline during first 12 weeks of treatment but stopped therapy due to inadequate virologic response iv. Relapse : Undetectable HCV RNA (HCV RNA <LLOQ) on treatment, but experienced breakthrough or relapse
* HIV-1 infection as documented by HIV-1 antibody at screening or any time prior to screening
* HIV treatment status: For subject receiving ART, HIV RNA must be < 40 copies/ml at screening and <200 copies/ml for at least 12 weeks prior to screening. Changes in therapy during the 12 weeks prior to enrollment permitted as long as not due to HIV treatment failure.
* HIV ART allowed in this study are the following and should be administered per the prescribing information in the package insert:

  * NRTIs: emtricitabine, lamivudine, tenofovir, abacavir
  * Maraviroc
  * Integrase inhibitors: dolutegravir or raltegravir
  * NNRTI's: rilpivirine
  * Enfuvitide Fixed dose combinations are permitted.
* Screening ECG without clinically significant abnormalities
* Subjects must have the following laboratory parameters at Screening and at Pre-entry (if pre-entry visit is required):

  * CD4 T-cell count >100 cells/mm3 if on ART, ≥ 350 cells/mm3 if not on ART
  * ALT ≤10 x the upper limit of normal (ULN)
  * AST ≤10 x ULN
  * Direct bilirubin ≤1.5 ULN
  * Creatinine clearance (CrClr) ≥50 mL /min, as calculated by the Cockcroft-Gault equation
  * Hemoglobin ≥10 g/dL
  * Albumin ≥3g/dL
  * INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
  * Alpha feto protein (AFP) levels <50. If ≥ 50, they should have a liver imaging study (eg, ultrasound, CT scan, MRI) showing no evidence of hepatocellular carcinoma within 3 months of study enrollment
* Female subjects of reproductive potential (defined as women who have not been post-menopausal for at least 24 consecutive months, ie, who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy) must have a negative serum pregnancy test with a sensitivity of at least 25 mIU/mL performed during screening, within 48 hours prior to study entry.
* All subjects must agree not to participate in a conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).

NOTE: Female candidates who are pregnant or breastfeeding are not eligible. A male candidate who has a pregnant female partner is not eligible for the study.

* When participating in sexual activity that could lead to pregnancy, all subjects must agree to use at least two non-hormonal forms of contraceptive simultaneously while receiving protocol-specified medications, and for 4 weeks after stopping the medications. Such methods include:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Tubal ligation NOTE: Providers and subjects should be advised that not all contraceptive choices listed above can prevent HIV transmission and that some may actually increase the risk of HIV acquisition. Study subjects who are sexually active with HIV-1 negative or unknown HIV-1 serostatus partners should be advised that they need to consider effective strategies for reducing the risk of HIV transmission, as well as meeting the requirement for effective contraception during their participation in the study. Study subjects should discuss contraceptive choices and HIV risk reduction methods with their health care provider.
* Subjects who are not of reproductive potential (women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy or men who have documented azoospermia or undergone vasectomy) are eligible without requiring the use of contraceptives. Acceptable documentation of sterilization and menopause is specified below.

Written or oral documentation communicated by clinician or clinician's staff of one of the following:

* Physician report/letter
* Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
* Discharge summary
* Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.

  * Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria:

* Hepatic decompensation at any point in time (includes variceal bleeding, hepatic encephalopathy, and ascites)
* HBs Ag +
* Prior HCV treatment with an HCV protease inhibitor or HCV polymerase inhibitor including sofosbuvir
* Other known causes of significant liver disease including chronic or acute hepatitis B, acute hepatitis A, hemochromatosis, or homozygote alpha-1 antitrypsin deficiency.
* Serious illness including malignancy within 24 weeks prior to study entry, or other chronic medical conditions that in the opinion of the site investigator may preclude completion of the protocol.
* Presence of active or acute AIDS-defining opportunistic infections within 12 weeks prior to study entry.
* Use of any prohibited concomitant medications
* Child-Pugh Score 6.2.2 Pre-entry>6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Estimated); Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
SVR12 (HCV RNA <LLOQ, or lower limit of quantification) | 12 weeks after discontinuation of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Luetkemeyer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Kirk GD, Mehta SH, Astemborski J, Galai N, Washington J, Higgins Y, Balagopal A, Thomas DL. HIV, age, and the severity of hepatitis C virus-related liver disease: a cohort study. Ann Intern Med. 2013 May 7;158(9):658-66. doi: 10.7326/0003-4819-158-9-201305070-00604. PMID 23440167
- [Background] Sulkowski MS, Mehta SH, Torbenson MS, Higgins Y, Brinkley SC, de Oca RM, Moore RD, Afdhal NH, Thomas DL. Rapid fibrosis progression among HIV/hepatitis C virus-co-infected adults. AIDS. 2007 Oct 18;21(16):2209-16. doi: 10.1097/QAD.0b013e3282f10de9. PMID 18090048
- [Background] Osinusi A, Meissner EG, Lee YJ, Bon D, Heytens L, Nelson A, Sneller M, Kohli A, Barrett L, Proschan M, Herrmann E, Shivakumar B, Gu W, Kwan R, Teferi G, Talwani R, Silk R, Kotb C, Wroblewski S, Fishbein D, Dewar R, Highbarger H, Zhang X, Kleiner D, Wood BJ, Chavez J, Symonds WT, Subramanian M, McHutchison J, Polis MA, Fauci AS, Masur H, Kottilil S. Sofosbuvir and ribavirin for hepatitis C genotype 1 in patients with unfavorable treatment characteristics: a randomized clinical trial. JAMA. 2013 Aug 28;310(8):804-11. doi: 10.1001/jama.2013.109309. PMID 23982366
- See also: Positive Health Program, San Francisco General Hospital/University of California, San Francisco — http://hiv.ucsf.edu/